CLINICAL TRIAL: NCT06337617
Title: A Multi-center Retrospective Study With Secondary Use of Data of Tafinlar (Dabrafenib) Plus Mekinist (Trametinib) in Chinese Patients With BRAF V600 Mutation Positive Melanoma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CDRB436B2407
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: BRAF V600 Mutation Positive Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort A (mucosal melanoma patients)
- Cohort B (non-mucosal melanoma patients)

SUMMARY:
This was a multi-center, observational, retrospective cohort study to evaluate the effectiveness and safety of dabrafenib in combination with trametinib in Chinese patients with unresectable or metastatic BRAF V600 mutation positive melanoma, for mucosal melanoma patients (Cohort A) and non-mucosal melanoma patients (Cohort B, cutaneous and acral melanoma), separately. Study population was identified as patients initiating dabrafenib plus trametinib from 01 May 2020 to 31 July 2022 who fulfilled the inclusion/exclusion criteria. The follow-up period ended at the earliest of the following: end of study observation period (i.e., 31 December 2022), death, upon withdrawal of consent or the last available record.

ELIGIBILITY:
Inclusion Criteria:

Cohorts A and B:

* Initiated dabrafenib and trametinib combination therapy (D+T) according to approved label between 01 May 2020 and 31 July 2022
* Was ≥18 years old of age at the initiation of D+T
* Had at least one tumor assessment after initiation of D+T
* Written informed consent if requested by the study site

Cohort A Only • Confirmed BRAF V600 mutation positive mucosal melanoma that was unresectable or metastatic

Cohort B Only

• Confirmed BRAF V600 mutation positive non-mucosal melanoma (cutaneous and acral melanoma) that was unresectable or metastatic

Exclusion Criteria:

None specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Real-world overall response rate (rwORR) | Up to approximately 2.6 years
  ORR was defined as the percentage of patients demonstrating a best overall response as complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or as documented per physician assessment, as available.

SECONDARY OUTCOMES:
Mean Age | Baseline
Percentage of patients per sex | Baseline
Number of years of disease history at treatment initiation since initial melanoma diagnosis | Baseline
Number and percentage of patients per anatomic sites of origin | Baseline
Number of years of disease history at treatment initiation since unresectable or metastatic melanoma diagnosis | Baseline
Number and percentage of patients per tumor stage | Baseline
Number and percentage of patients with occurrence of tumor metastasis | Baseline
Number and percentage of patients per metastatic location | Baseline
Number and percentage of patients per metastases | Baseline
Lactate dehydrogenase (LDH) levels | Baseline
Eastern Cooperative Oncology Group (ECOG) performance status | Baseline
  ECOG performance status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scores can range from a lower value of 0 (fully active, able to carry on all pre-disease performance without restriction) up to 5 (dead).
Number and percentage of patients who had at least one surgery for melanoma prior to D+T treatment | Baseline
Number and percentage of patients per type of surgery | Baseline
Number and percentage of patients per name of surgery | Baseline
Number and percentage of patients per surgical and medical procedure | Baseline
Number and percentage of patients who had at least one anti-neoplastic drug for melanoma prior to D+T treatment | Baseline
Number and percentage of patients with prior anti-neoplastic drugs for melanoma per treatment intent | Baseline
Number and percentage of patients with prior anti-neoplastic drug for melanoma per treatment setting | Baseline
Number and percentage of patients with prior anti-neoplastic drug for melanoma per line of treatment | Baseline
Number and percentage of patients with prior anti-neoplastic drug for melanoma per treatment type | Baseline
Number and percentage of patients per reason for immunotherapy discontinuation | Baseline
Number and percentage of patients with prior anti-neoplastic drug for melanoma with best overall tumor response | Baseline
Number and percentage of patients per prior anti-neoplastic drug for melanoma | Baseline
Number and percentage of patients who had at least one radiotherapy for melanoma prior to D+T treatment | Baseline
Number and percentage of patients with prior radiotherapy for melanoma per treatment intent | Baseline
Number and percentage of patients with prior radiotherapy for melanoma per treatment setting | Baseline
Number and percentage of patients per radiation site | Baseline
Mean total dosage for all radiotherapy | Baseline
Number and percentage of patients with prior radiotherapy for melanoma with best overall tumor response | Baseline
Number and percentage of patients with dabrafenib plus trametinib treatment per line of treatment | Up to approximately 2.2 years
Number and percentage of patients with dabrafenib plus trametinib treatment per treatment intent | Up to approximately 2.2 years
Number and percentage of patients with dabrafenib plus trametinib treatment per treatment setting | Up to approximately 2.2 years
Number and percentage of patients per type of D+T treatment change | Up to approximately 2.2 years
Number and percentage of patients per reason for D+T treatment change | Up to approximately 2.2 years
Mean duration of D+T, if not ongoing to end of study follow-up | Up to approximately 2.2 years
rwORR of dabrafenib plus trametinib among non-mucosal melanoma patients (FAS) | Up to approximately 2.6 years
Real-world disease control rate (rwDCR) of D+T (FAS) | Up to approximately 2.6 years
  rwDCR was defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) or non-CR or non-progressive disease (non-PD), per RECIST version 1.1 or as documented per physician assessment, as available.
Real-world duration of response (rwDOR) of dabrafenib plus trametinib | Up to approximately 2.6 years
  For the subset of patients with CR or PR, rwDORn was defined as the time from the date of the first documented CR or PR per RECIST version 1.1 or as documented per physician assessment as available, to the first disease progression or death due to any cause.
Real-world progression-free survival (rwPFS) for dabrafenib plus trametinib (FAS) | Up to approximately 2.6 years
  rwPFS was defined as the time from the start of treatment to the first documented disease progression or death due to any cause.
Real-world overall survival (rwOS) since D+T initiation (FAS) | Up to approximately 2.6 years
  rwOS was defined as the time from start of treatment to death due to any cause.
Time to treatment discontinuation (FAS) | Up to approximately 2.6 years
Number and percentage of patients with adverse events of special interest (AESIs) (FAS) | Up to approximately 2.6 years
  AESIs were defined based on the case retrieval strategy file available at the time of analysis.
Number and percentage of patients with serious adverse events (SAEs) (FAS) | Up to approximately 2.6 years
rwPFS for dabrafenib plus trametinib (MMS), by immunotherapy use | Up to approximately 2.6 years
  rwPFS was defined as the time from the start of treatment to the first documented disease progression or death due to any cause.
rwPFS for dabrafenib plus trametinib (NMS), by immunotherapy use | Up to approximately 2.6 years
  rwPFS was defined as the time from the start of treatment to the first documented disease progression or death due to any cause.
rwOS since D+T initiation (MMS), by immunotherapy use | Up to approximately 2.6 years
  rwOS was defined as the time from start of treatment to death due to any cause.
rwOS since D+T initiation (NMS), by immunotherapy use | Up to approximately 2.6 years
  rwOS was defined as the time from start of treatment to death due to any cause.
Number and percentage of patients with systemic anti-neoplastic treatment after D+T | Up to approximately 2.6 years
Number and percentage of patients with systemic anti-neoplastic treatment after D+T per line of treatment | Up to approximately 2.6 years
Number and percentage of patients with systemic anti-neoplastic treatment after D+T and treatment ongoing at end of follow up | Up to approximately 2.6 years
Number and percentage of patients with systemic anti-neoplastic treatment after D+T per treatment type | Up to approximately 2.6 years
Number and percentage of patients per reason for immunotherapy discontinuation | Up to approximately 2.6 years
Number and percentage of patients with systemic anti-neoplastic treatment after D+T with best overall tumor response | Up to approximately 2.6 years
Number and percentage of patients who had systemic anti-neoplastic treatment after D+T treatment | Up to approximately 2.6 years
Number and percentage of patients who had systemic anti-neoplastic treatment after D+T treatment per medication | Up to approximately 2.6 years
Number and percentage of patients per concomitant medication | Up to approximately 2.2 years
Real-world overall survival since the first anti-neoplastic drug treatment for advanced/metastatic melanoma (FAS) | Up to approximately 2.6 years
Real-world overall survival since the first anti-neoplastic drug for advanced/metastatic melanoma (NMS), by immunotherapy use | Up to approximately 2.6 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Shanghai, China